CLINICAL TRIAL: NCT04209010
Title: Comparison of One-stage Direct-to-implant With Acellular Dermal Matrix and Two-stage Implant-based Breast Reconstruction: A Cohort Study
Brief Title: Immediate Breast Reconstruction With Acellular Dermal Matrix
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Cancer Society (Other); The Korning foundation (Unknown); Foundation of the Kjaersgaard Family (Unknown); King Christian X foundation (Unknown); Foundation of architect Holger Hjortenberg (Unknown); LifeCell Corporation (Branchburg, NJ, USA) (Unknown)
Responsible Party: Principal Investigator, Mette Eline Brunbjerg, MD, MD, PhD student, Principal Investigator, Aarhus University Hospital
Other Study IDs: VEK 1-10-72-572-12
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Breast Carcinoma in Situ; Mammaplasty; Acellular Dermis
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- One-stage group: Immediate implant based breast reconstruction after skin sparing mastectomy in one stage using silicone implant and acellular dermal matrix.
  Interventions: Procedure: one-stage technique
- Two-stage group: Immediate implant based breast reconstruction after skin sparing mastectomy in two stages using expander to silicone implant technique.

INTERVENTIONS:
Procedure: one-stage technique — breast reconstruction in one stage using silicone implant and acellular dermal matrix.
  Groups: One-stage group

SUMMARY:
The aim of this study is to contribute to the knowledge regarding immediate implant-based BR by investigating whether the one-stage technique with ADM is superior to the two-stage expander to implant technique. Primary endpoint in first publication is postoperative complications, secondary endpoint is patient and investigator assessed aesthetic outcome. Primary endpoint in second publication is cost, secondary endpoint is patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Skin sparing mastectomy due to breast cancer, ductal carcinoma in situ or high genetic risk of developing breast cancer
* Mastectomy weight ≤ 600 g
* Patient older than 18 years
* Ability to complete the study questionnaire
* Only for the two-stage group no later than 2 years and 4 months from breast reconstruction

Exclusion Criteria:

- smokers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were all women admitted for immediate, implant-based breast reconstruction following skin-sparing mastectomy at the Department of Plastic and Breast Surgery, Aarhus University Hospital, Denmark from September 2010 to January 2014.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 3 months
  Major (requiring surgery - infection, hematoma, mastectomy flap necrosis). Obtained by review of patient chart.
Postoperative complications | 3 months
  Minor (not requiring surgery - seroma, cellulitis). Obtained by review of patient chart.

SECONDARY OUTCOMES:
Patient assessed satisfaction with aesthetic result | 2 years
  Assessment of result with and without clothes, symmetry and all-in-all satisfaction with result. Obtained by questionnaire on a 7 point Likert scale. Higher score equals higher satisfaction.
Investigator assessed satisfaction with aesthetic result | 2 years
  Assessment of result with and without clothes, symmetry (including measurements of sternal notch-papil distance and papilla-inframammary fold distance). Obtained by clinical examination.
Patient reported outcome measures | 2 years
  Patient reported assessment of pain and dysaesthesia in reconstructed breast, arm/shoulder function on reconstructed side. Described on a 6 point scale where lower score equals more pain/dysaesthesia/troubles with arm/shoulder function.
  Body image (Hopwoods Body Image Scale) assessed in a 10-items each on 4 point Likert scale from 0 to 3. Sum provides a total score (range 0-30) and lower scores equals less body image troubles.
  Furthermore, study specific questions as "use of pain killers the last week" (yes / no) and "all in all assessment of health owning to the breast reconstruction" (improved / diminished or unchanged). All obtained by questionnaire.
Cost | 2 years
  cost analysis comparing the two methods regarding hospitalization, out patient visits, cost of expander/implant/acellular dermal matrix, surgical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Eline Brunbjerg, MD, Principal Investigator — Aarhus University Hospital, Aarhus University, Denmark

IPD SHARING:
Plan to Share IPD: No
All data will be anonymized.

REFERENCES:
- [Derived] Brunbjerg ME, Jensen TB, Overgaard J, Christiansen P, Damsgaard TE. Comparison of one-stage direct-to-implant with acellular dermal matrix and two-stage immediate implant-based breast reconstruction-a cohort study. Gland Surg. 2021 Jan;10(1):207-218. doi: 10.21037/gs-20-581. PMID 33633977